CLINICAL TRIAL: NCT01585818
Title: Nutrition Studies and Dietary Intervention in Individuals With Type 2 Diabetes Mellitus of Chinese, Malay and Indian Ethnicity
Brief Title: Dietary Intervention in Diabetes Mellitus (DIDM)- Intermediate and Acute Effects
Acronym: DIDM
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Collaborators: National Medical Research Council (NMRC), Singapore (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SICS-10/1/2/002
Record Dates: First submitted 2012-04-25; First posted 2012-04-26 (Estimated); Last update posted 2014-01-17 (Estimated); Status verified 2014-01

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Glycemic Index; Type 2 Diabetes Mellitus; Diet; Glucose Variability; Metabolic Response; Glucose Response
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- standard dietary intervention (SDI) arm (Active Comparator): The general principles for the SDI arm are to provide an understanding of carbohydrates, be isocaloric based on assessment from the food diary/ recall and anthropometric measures, provide a personalised even distribution of carbohydrate throughout the day, have general recommendations such as reduction of fat, sodium, sugar and an increase in fibre
  Interventions: Other: Standard Diet Intervention
- LGI intervention arm (Experimental): The general principles for the LGI intervention arm include the SDI principles and instructions on GI, identifying foods of different GI, switching to low GI food and having at least one low GI food per meal and suggested meals with recipes. Participants will also have the opportunity to attend sessions to learn how to cook meals with low GI. Participants will be provided with a list of low GI carbohydrates to consume during the intervention period and in addition, they will be provided with a supply of the staples for the same period
  Interventions: Other: Low Glycemic Index (LGI) intervention arm

INTERVENTIONS:
Other: Low Glycemic Index (LGI) intervention arm — The general principles for the LGI intervention arm include the SDI principles and instructions on GI, identifying foods of different GI, switching to low GI food and having at least one low GI food per meal and suggested meals with recipes. Participants will also have the opportunity to attend sessions to learn how to cook meals with low GI.
  Other Names: Low GI
  Arms: LGI intervention arm
Other: Standard Diet Intervention — The general principles for the SDI arm are to provide an understanding of carbohydrates, be isocaloric based on assessment from the food diary/ recall and anthropometric measures, provide a personalised even distribution of carbohydrate throughout the day, have general recommendations such as reduction of fat, sodium, sugar and an increase in fibre. Participants will be provided with a list of carbohydrates to take during the intervention period and will be provided a supply of carbohydrates for that period
  Other Names: SDI arm
  Arms: standard dietary intervention (SDI) arm

SUMMARY:
Lifestyle modification, in particular adopting an appropriate dietary pattern, is generally accepted as the cornerstone for the treatment of people with type 2 diabetes mellitus (T2DM). Consumption of low glycaemic index (GI) meals have been shown to improve glycaemic control, lipid profile and reduced systemic inflammation. However, these studies and international evidence-based nutritional recommendations are principally based on people of European ethnicity consuming fairly typical "western" diets. There are few published controlled dietary intervention studies which have attempted to determine appropriate dietary patterns for the treatment of diabetes amongst populations consuming rice-based diets.

HYPOTHESIS

1. The glycaemic response over 6 days as measured by CGMS will have a lower mean glucose level and postprandial increase in individuals consuming the LGI compared with the SDI meal plan.
2. A LGI meal plan is acceptable and participants will adhere and comply to the diet to the same level as those receiving the SDI meal plan.
3. Glycaemic and metabolic parameters as measured by integrated area under the curve (IAUC) of glucose and insulin are lower after a single meal comprising of LGI than compared with an SDI meal.
4. The effect of a single meal of LGI reduces appetite and increases satiety compared with a meal of SDI.

DETAILED DESCRIPTION:
This study builds on the information collected from phase 1 which involved the documentation of clinical and metabolic characteristics and dietary practices of Chinese individuals with T2DM. In addition to information from a separate study on GI testing of locally consumed carbohydrate containing foods, we have formulated a meal plan comprising of low GI carbohydrates. Participants will be randomised into the low GI (LGI) intervention arm or standard dietary intervention (SDI) arm and receive counselling and advice from a dietitian, embark on a two week protocol to test the recommended diet, be reviewed by the dietitian, and undergo a 3 to 6 day continuous glucose monitoring period before and after the LGI or SDI diet. In addition, they will undergo 2 separate single day test meals comprising of low GI and high GI foods. Participants in both groups will be given resources including detailed instructions and meal plans that are comparable between the two arms in terms of contact with research personnel, instructions and meal plans which are isocaloric and have similar macronutrient composition appropriate for their energy requirements.

Participants will be advised to continue on the meal plans and diet for a further 22 weeks. At the second month, a telephone call will be made to the participant to review compliance. At month 3 and month 6, participants will be asked to attend after an overnight fast from 10pm, for a blood sample, return a food diary/ recall, measurement of anthropometry and blood pressure. In addition, they will complete a questionnaire

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to comply with study procedures and give written informed consent
2. Have established diagnosis of type 2 diabetes* of more than 1 year on diet treatment or oral anti-diabetic therapy
3. Male or female, aged 45 to 64 years inclusive
4. HbA1c of 7.0 - 10.0% (inclusive) within the last 3 months or at screening
5. Stable glycaemic control
6. Patients with concurrent illnesses if medically stable for 6 months prior to screening visit, based on the clinical judgement of the investigator
7. Be on stable therapy (no significant change to therapy in last 3 months)
8. No hospitalization or surgery in the past 6 months
9. No use of corticosteroids in the last 6 months
10. Not pregnant
11. Urea <30 mmol/L and estimated GFR >= 60ml/min
12. Be willing to prepare and adhere to the meal plans and consume at least two meals at home per day.
13. Be willing and able to undertake blood glucose monitoring, continuous glucose monitoring.

    * Subjects with Type 2 DM should have been diagnosed at least 1 years prior to the screening visit and should not have T1DM, MODY or secondary diabetes e.g. diabetes secondary to chronic pancreatitis

Exclusion Criteria:

1. Significant medical conditions which in the Investigator's opinion would confound interpretation of the results, including but not limited to: current symptomatic cardiovascular disease, macroalbuminuria (dipstick positive proteinuria on more than 1 consecutive occasion) or renal impairment (serum creatinine above 120 umol/l), cancer, overt liver disease other than Non Alcoholic Steatohepatitis (liver enzyme levels less than 3 times upper limit of normal) or gastroparesis.
2. Recent changes in weight of >5% over the past 6 months
3. Significant changes in diet over the past 6 months
4. Any use of weight reducing drugs, or on medications such as alpha-glucosidase inhibitors or insulin currently or in the past 6 months
5. Any surgery (and bariatric surgery) in the past 6 months
6. Any use of investigational drugs in the past 6 months
7. Any serious illness requiring hospitalization in the past 6 months
8. Any use of corticosteroids in the past 6 months
9. Ongoing infection, or condition that interfered with nutrient digestion, absorption, metabolism or excretion (including gastroparesis)
10. Allergy or intolerant to the ingredients or any of the food items in the intervention diet or to paracetamol/ acetaminophen

Ages: 45 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2011-08; Primary Completion 2014-05 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Average mean glucose levels and variability | 2 weeks
  To assess the intermediate effects on glycaemia and metabolic response to a meal plan comprising of LGI compared with a SDI meal plan

SECONDARY OUTCOMES:
HBA1C | 3 and 6 months
  1. To assess acceptability and compliance to the intervention meal plan
  2. To assess the intermediate effects of glycaemia
Glucose and Insulin Levels | 1 week
  To assess glycemic and metabolic response to a mixed meal

CONTACTS AND LOCATIONS:
Overall Officials: Eric YH Khoo, MD, Principal Investigator — National University Hospital / Medicine
Locations (1):
- National University Hospital, Singapore, Singapore